CLINICAL TRIAL: NCT01428713
Title: Prospective Crossover Trial of Oral Tranexamic Acid and Combined Oral Contraceptive in Adolescents With Menorrhagia - A Pilot Study
Brief Title: Tranexamic Acid (TA) vs Combined Oral Contraceptive (COCP) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Lakshmi Srivaths, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-27934 TA vs COCP Study
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Menorrhagia
Keywords: menorrhagia; oral contraceptives; oral tranexamic acid
MeSH Terms: conditions — Menorrhagia | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A-Oral tranexamic acid (Active Comparator): Group A received oral tranexamic acid at 1300 mg (two 650mg tablets), three times each day on days 1 to 5 of menstrual cycle for 3 cycles.
  Interventions: Drug: Oral tranexamic acid
- Group B-Combined oral contraceptive pills (Active Comparator): Group B received combined oral contraceptive pills with 3 weeks of hormonal pills and 1 week of placebo for 3 cycles.
  Interventions: Drug: Oral Contraceptive Pills

INTERVENTIONS:
Drug: Oral tranexamic acid — Group A received oral tranexamic acid at 1300 mg (two 650mg tablets), three times each day on days 1 to 5 of menstrual cycle for 3 cycles.
  Arms: Group A-Oral tranexamic acid
Drug: Oral Contraceptive Pills — Group B received combined oral contraceptive pills with 3 weeks of hormonal pills and 1 week of placebo for 3 cycles.
  Arms: Group B-Combined oral contraceptive pills

SUMMARY:
Menorrhagia, considered a public health challenge and reported by 5 to 10% of adult women, is encountered even more frequently in adolescents. Surveys of school students in the United States (US) and Europe reported menorrhagia in 37% to 55% of adolescent females. Medical management of adolescent menorrhagia includes various formulations of hormonal therapy and the antifibrinolytic agent epsilon aminocaproic acid. Oral tranexamic acid (TA), a more potent antifibrinolytic agent used as standard therapy for menorrhagia in adult women and in adolescent women in Europe and Canada, was not previously available in the US. Subsequent to US FDA approval in November 2009 of a novel oral TA formulation to treat cyclic heavy menstrual bleeding in adult women, this medication is currently included in the treatment armamentarium for adult menorrhagia. There is currently no preliminary data available in the US about the clinical use of oral TA in an exclusive adolescent population with menorrhagia. Oral contraceptive pills (OCP) are considered standard therapy in the management of menorrhagia in teen-aged women. Oral TA has been shown to be more efficacious than progesterone-only hormonal therapy for menorrhagia in adult women. However, there is no data available comparing the efficacy of oral TA and combined OCP (COCP) in adult women or in adolescents with menorrhagia.

The study hypothesis is that, in adolescent menorrhagia, oral TA will have comparable efficacy in reducing menstrual blood loss (MBL) and improving quality of life (QOL) when compared to the commonly prescribed COCP.

This hypothesis was tested by comparing the efficacy of these two medications, in a prospective randomized crossover trial in post-menarchal young girls with menorrhagia.

DETAILED DESCRIPTION:
Subjects were randomized to one of two groups (group A or B).

Group A received oral tranexamic acid at 1300 mg (two 650mg tablets), three times each day on days 1 to 5 of menstrual cycle for 3 cycles.

Group B received combined oral contraceptive pills (OCP) with 3 weeks of hormonal pills and 1 week of placebo for 3 cycles.

After 3 cycles of therapy, both groups had one cycle without any therapy. Then, the groups crossed over. Group A, who first received TA, then received OCP. Group B, who first received OCP, then received TA.

All subjects were to receive both tranexamic acid and oral contraceptive pills.

There were a total of 3 study-associated visits per patient: 1 at baseline and 2 at the end of 3 cycles on each medication. These visits were considered within standard of care, as subjects with menorrhagia have frequent monitoring until the effectiveness of the treatment is determined.

At the study visits the following were done:

1. Assessment of the last menstrual period (amount of blood lost) using the Pictorial Blood Assessment Chart (PBAC) score and the number of days the period lasted
2. Quality of Life evaluation - by the patient completing a standardized pediatric quality of life (PedsQL) questionnaire
3. Detailed history and physical examination to evaluate for drug side effects and to look for signs of blood clots.
4. Blood drawn for a complete blood count.

ELIGIBILITY:
Inclusion Criteria:

1. Menstruating females with menorrhagia or menometrorrhagia referred to hematology or gynecology clinics at Texas Childrens Hospital. Menorrhagia is defined as regular periods with heavy menstrual bleeding with a PBAC score greater than 100; menometrorrhagia is heavy vaginal bleeding occurring at irregular intervals.
2. PBAC Score greater than 100 for 2 consecutive cycles
3. Pelvic ultrasound that excludes pelvic pathology that can cause menorrhagia within 12 months prior to study participation.
4. Normal external genitalia examination within 6 months prior to study participation.
5. Normal thyroid stimulating hormone (TSH) in the last 6 months prior to study participation.
6. Negative urine or serum pregnancy test within 4 weeks prior to study participation.

Exclusion Criteria:

1. Presence of intra uterine device.
2. Presence of a diagnosed bleeding disorder based on the standard work-up including complete blood count (CBC), prothrombin time, partial thromboplastin time, fibrinogen, von Willebrand panel and platelet function analysis (PFA-100) or platelet aggregation.
3. Intake of medications with increased risk of bleeding
4. Taking herbal products.
5. Sexually active status.
6. Body weight less than 40 kg.

Max Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Srivaths, MD, Principal Investigator — Baylor College of Medicine/TCH
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post-menarchal young girls </= 21 years of age with menorrhagia or menometrorrhagia, referred to hematology or gynecology clinics at Texas Children's Hospital (TCH) formed the study population.
Pre-assignment Details: The study design employed was a randomized crossover trial comparing the use of oral TA formulation Lysteda and the COCP formulation Lo/Ovral. Patients were randomized to one of two treatment groups, group A versus group B. Patients who were already on COCP underwent one cycle washout prior to randomization.
Groups:
- Group A: TA First, Then COCP: Patients received oral TA (given according to US FDA label for adult women, an off-label use for adolescents <18 years of age) at 1300 mg (two 650mg tablets) three times each day on days 1 to 5 of menstrual cycle for 3 consecutive cycles.
  Subsequently, patients who initially received TA, received COCP. COCP formulation Lo/Ovral (components: Ethinyl estradiol 30 mcg and norgestrel 0.3 mg; each monthly pack containing 21 hormonal tablets and 7 inactive tablets). Patients received COCP with 3 weeks of hormonal pills and 1 week of placebo pills for 3 consecutive cycles. Each medication was prescribed for 3 menstrual cycles with a 1 month wash out in-between TA and COCP.
- Group B: COCP First, Then TA: Patients received COCP first. COCP formulation Lo/Ovral (components: Ethinyl estradiol 30 mcg and norgestrel 0.3 mg; each monthly pack containing 21 hormonal tablets and 7 inactive tablets). Patients received COCP with 3 weeks of hormonal pills and 1 week of placebo pills for 3 consecutive cycles. Each medication was prescribed for 3 menstrual cycles with a 1 month wash out in-between COCP and TA.
  Subsequently, patients who initially received COCP, received TA. Patients received oral TA (given according to US FDA label for adult women, an off-label use for adolescents <18 years of age) at 1300 mg (two 650mg tablets) three times each day on days 1 to 5 of menstrual cycle for 3 consecutive cycles.
Period: Overall Study
Arm/Group | Group A: TA First, Then COCP | Group B: COCP First, Then TA
Started | 9 | 8
Completed | 6 | 3
Not Completed | 3 | 5
Not completed — Non-compliance | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: 17 post-menarchal girls with menorrhagia or menometrorrhagia without underlying bleeding disorders, pelvic pathology, pelvic infection, thyroid abnormalities or pregnancy.
Groups:
- All Study Participants: Group A: TA first, then COCP:
  Patients received oral TA (given according to US FDA label for adult women, an off-label use for adolescents <18 years of age) at 1300 mg (two 650mg tablets) three times each day on days 1 to 5 of menstrual cycle for 3 consecutive cycles.
  Subsequently, patients who initially received TA, received COCP.
  Group B: COCP first, then TA:
  Patients received COCP first. COCP formulation Lo/Ovral (components: Ethinyl estradiol 30 mcg and norgestrel 0.3 mg; each monthly pack containing 21 hormonal tablets and 7 inactive tablets). Patients received COCP with 3 weeks of hormonal pills and 1 week of placebo pills for 3 consecutive cycles. Each medication was prescribed for 3 menstrual cycles with a 1 month wash out in-between TA and COCP.
  Subsequently, patients who initially received COCP, received TA.
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Continuous [Median (Standard Deviation); unit: years] | 14.2 (1.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: To Assess the Efficacy of Oral TA and COCP in Adolescents With Menorrhagia.
Description: To assess
  1. change in Pictorial Blood Assessment Chart Score (PBAC Score) from baseline to the end of 3 cycles of TA
  2. change in quality of life (QOL) as evaluated by the PedsQL instrument from baseline to the end of 3 cycles of TA
  3. change in Pictorial Blood Assessment Chart Score (PBAC Score) from baseline to the end of 3 cycles of COCP
  4. change in quality of life (QOL) as evaluated by the PedsQL instrument from baseline to the end of 3 cycles of COCP
  PBAC score:
  Quantitative score to measure menstrual blood loss. Scale range: Minimum - 0 score, Maximum: No maximum Interpretation: Score > 100 indicates heavy menstrual bleeding
  Peds QL score:
  Score to measure quality of life in children Scale range: Minimum: 0, Maximum 100 Calculation: Subscales are reverse scored (using formula 100 - a x 25) and then all subscales are averaged Eg: Subscale score of 3 is reverse scored as: 100 - (3 x 25) = 25 Interpretation: Higher score indicates better quality of life
Time Frame: Baseline, 3 cycles
Population: 10 patients completed TA and their results were analyzed. 11 patients completed COCP and their results were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Group: TA: Patients received oral TA (given according to US FDA label for adult women, an off-label use for adolescents <18 years of age) at 1300 mg (two 650mg tablets) three times each day on days 1 to 5 of menstrual cycle for 3 consecutive cycles.
- Group: COCP: Patients received COCP formulation Lo/Ovral (components: Ethinyl estradiol 30 mcg and norgestrel 0.3 mg; each monthly pack containing 21 hormonal tablets and 7 inactive tablets). Patients received COCP with 3 weeks of hormonal pills and 1 week of placebo pills for 3 consecutive cycles.
Arm/Group | Group: TA | Group: COCP
Number analyzed (Participants) | 10 | 11
Scores on a scale
  PBAC (Pictorial Blood Assessment Chart) score | 536.4 (162.12) | 430.6 (157.35)
  Peds QL (Pediatric Quality of Life) score | 15.6 (5.08) | 16.75 (4.87)
Statistical Analysis 1: Comparison: Group: TA; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis — P value < 0.05 is considered significant in this study; Mean Difference (Final Values) = 536.4, Standard Error of Mean 162.12 — Comparing PBAC score value at baseline vs. end of 3 cycles for TA
Statistical Analysis 2: Comparison: Group: COCP; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — P value < 0.05 is considered significant for this study; Mean Difference (Final Values) = 430.6, Standard Error of Mean 157.35 — Comparing PBAC score value at baseline vs. end of 3 cycles for COCP
Statistical Analysis 3: Comparison: Group: TA; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis — P value < 0.05 is considered significant for this study; Mean Difference (Final Values) = 15.6, Standard Error of Mean 5.08 — Comparing Peds QL score value at baseline vs. end of 3 cycles for TA
Statistical Analysis 4: Comparison: Group: COCP; Test type: Superiority or Other; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 16.75, Standard Error of Mean 4.87 — Comparing Peds QL score value at baseline vs. end of 3 cycles for COCP

ADVERSE EVENTS:
Time Frame: 8 months
Description: Only patients that completed each intervention were considered at risk. 10 patients completed TA and their results were analyzed. 11 patients completed COCP and their results were analyzed.
Groups:
- Tranexamic Acid (TA): Patients received oral tranexamic acid at 1300 mg three times each day on days 1 to 5 of menstrual cycle for 3 cycles. The mean age of the study population was 14.2 years. Patients received oral TA (given according to US FDA label for adult women, an off-label use for adolescents <18 years of age) at 1300 mg (two 650mg tablets) three times each day on days 1 to 5 of menstrual cycle for 3 consecutive cycles.
  Subsequently, patients who initially received TA, received COCP and patients who initially received COCP, then received TA.
- Combined Oral Contraceptives (COCP): COCP formulation Lo/Ovral (components: Ethinyl estradiol 30 mcg and norgestrel 0.3 mg; each monthly pack containing 21 hormonal tablets and 7 inactive tablets). Patients received COCP with 3 weeks of hormonal pills and 1 week of placebo pills for 3 consecutive cycles. Each medication was prescribed for 3 menstrual cycles with a 1 month wash out in-between medications.
Arm/Group | Tranexamic Acid (TA) | Combined Oral Contraceptives (COCP)
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 2/10 | 8/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (TA) (N=10) | Combined Oral Contraceptives (COCP) (N=11)
breakthrough bleeding (Reproductive system and breast disorders) | 1 (1) | 1 (1)
nausea/vomiting (General disorders) | 1 (1) | 1 (1)
abdominal pain (General disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
weight gain (General disorders) | 0 (0) | 1 (1)
mood swings (General disorders) | 0 (0) | 1 (1)
depression and seizure (General disorders) | 0 (0) | 1 (1) — Depression and seizure already diagnosed prior to study.
generalized rash (General disorders) | 0 (0) | 1 (1)
Lack of sleep (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No